CLINICAL TRIAL: NCT04011683
Title: Hypoglycaemia and Cardiac Arrhythmias in Type 1 Diabetes
Acronym: Hypo-Heart-1
Status: Completed | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other); University Hospital, Gentofte, Copenhagen (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: H-18034040_part2
Record Dates: First submitted 2019-06-17; First posted 2019-07-08 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Hypoglycemia (Diabetic); Hyperglycaemia (Diabetic); Arrythmia, Cardiac; Type 1 Diabetes; Blood Glucose Fluctuations
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia; Arrhythmias, Cardiac; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators hypothesise that patients with type 1 diabetes have clinically relevant, but often unrecognised, episodes of arrhythmias linked to episodes of hypoglycaemia and/or clinically significant fluctuations in plasma glucose.

DETAILED DESCRIPTION:
30 patients with type 1 diabetes will be recruited for a one-year observational study employing CGM (Continuous glucose monitor) and ILR (Implantable loop recorder). Patients will be scheduled for a three-week run-in period to ensure that the implanted ILR provides reliable data. Patient visits are planned for 0, 3, 6, 9, and 12 months and will include clinical examination, blood and urine samples, echocardiography (only first and last visit) and implant/explant of CGM. After 12 months, the participants will continue with an extended observation period of 2 years employing ILR and clinical examination.

Device: Loop recorder (Reveal LINQ, Medtronic, Minneapolis, MN, USA) Implantation of a loop-recorder

Device: Continuous glucose monitoring (Eversense XL, Senseonics, USA) Monitoring with a continuous glucose monitor

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Type 1 diabetes diagnosed according to the criteria of the World Health Organization (WHO)
* Age 18-80 years
* Fulfilling at least one of the below criteria*:

  1. Recurrent hypoglycaemia (defined as >1 episode/week with a plasma glucose measurement ≤3.9 mmol/l within the last 4 weeks)
  2. An episode of severe hypoglycaemia within the last year (according to the ADA definition, an event requiring assistance of another person to actively administer carbohydrates and/or glucagon, or take other corrective actions)
  3. Hypoglycaemic symptom unawareness (history of impaired autonomic response during hypoglycaemia)

(*The aim is that all patients will fulfil criteria a or b. If the targeted sample size cannot be recruited, patients fulfilling criteria c will be included)

* Insulin treatment
* One or more clinical relevant complications to diabetes defined as**:

  1. Nephropathy (creatinine >130 μmol/l and/or microalbuminuria)
  2. Macrovascular disease defined as coronary disease (stable angina pectoris. previous unstable angina pectoris or myocardial infarction), cerebrovascular disease (previous stroke or transitional cerebral ischaemia), and peripheral vascular disease (previous intermittent claudication or prior acute ischemia)
  3. Peripheral neuropathy with vibration perception threshold of >25 volt determined by biothesiometry
  4. Moderate to severe retinopathy
* Well-functioning ILR during run-in period (acceptable readings judged by an arrhythmologist)
* Participation in the extended study

(**The aim is that all patients will fulfil criteria a or b. If the targeted sample size cannot be recruited, patients fulfilling criteria c or d will be included)

Exclusion Criteria:

* Arrhythmia diagnosed prior to the screening visit
* ICD or pacemaker at the time of inclusion
* Severe heart failure (left ventricular ejection fraction <25%)
* Structural heart disease (Wolf-Parkinson-White syndrome, congenital heart disease, severe valve disease)
* Thyroid dysfunction (except for well-regulated eltroxine substituted myxoedema)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 Diabetes recrutted in collaboration with Hillerod hospital, Gentofte hospital and Steno Diabetes Centre.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiac arrhythmias during hypoglycaemia, euglycaemia, hyperglycaemia. | Within 12 months
  Incidence of clinically relevant arrhythmias during hypoglycaemia (plasma glucose ≤3.9 mmol/l) compared to euglycaemia and hyperglycaemia.

SECONDARY OUTCOMES:
Prevalence of cardiac arrhythmias | Within 12 months
  Prevalence of clinically relevant arrhythmias
Cardiac arrhythmias during LGV, HGV. | Within 12 months
  Clinical relevant arrhythmias during low glucose variability (LGV), defined as variations in plasma glucose below or equal to 5 mmol/l within two hours preceding an arrhythmic event, compared to high glucose variability (HGV), defined as variations in plasma glucose above 5 mmol/l within two hours preceding an arrhythmic event.
The relationship between cardiovascular disease at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV | Within 12 months
  The relationship between cardiovascular disease (heart failure and ischaemic heart disease) at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV
The relationship between pharmacological treatment at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV | Within 12 months
  The relationship between pharmacological treatment at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV
The relationship between diabetes complication status at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV | Within 12 months
  The relationship between diabetes complication status (neuropathy, nephropathy, retinopathy) at baseline and clinically relevant arrhythmias in relation to hypoglycaemia and HGV
Hypoglycaemia and cardiac arrhythmia | Within 12 months
  The correlation between prevalence and total duration of hypoglycaemia and risk of clinically relevant arrhythmias
Plasma glucose variation and cardiac arrhythmias | Within 12 months
  The correlation between plasma glucose variation (variation in plasma glucose (Δ mmol/l) within two hours of the event) and risk of clinically relevant arrhythmias
CV, SD, ADRR, LBGI, HBGI, CONGA-1 and cardiac arrhythmias | Within 12 months
  The correlation between measures of glycaemic variability (coefficient of variation (CV), standard deviation (SD), average daily risk range (ADRR), low blood glucose index (LBGI), high blood glucose index (HBGI) and continuous overlapping net glycaemic action (CONGA-1)) and risk of clinically relevant arrhythmias
Mean amplitude of glycaemic excursions (MAGE) and cardiac arrhythmia. | Within 12 months
  Difference in mean amplitude of glycaemic excursions (MAGE) two hours preceding an arrhythmic event versus MAGE during non-event

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, MD, Professor, Study Director — Steno Diabetes Center Copenhagen
Locations (1):
- Clinical Metabolic Physiology, SDCC, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided